CLINICAL TRIAL: NCT07163260
Title: Defeat Rare Disease in Asia and Pacific (APAC) DRDA - Haemophilia
Status: Enrolling by invitation | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: DAS-8107; U1111-1303-7372 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-08-06; First posted 2025-09-09 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Haemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Experienced/Senior Treating Physicians: This group includes haematologists, paediatric haematologist and physicians treating patients with haemophilia (PWH)
  Interventions: Other: No treatment given
- Patients Organisations: This group includes the organisations working closely to support patient with haemophillia (PWH) at a national/regional level
  Interventions: Other: No treatment given
- Patients/Caregivers: This group includes patients with haemophilia and caregivers managing patients with haemophilia
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given

SUMMARY:
This study will help to better understand the course of disease in people with haemophilia (A or B [with or without inhibitors]) and the haemophilia care scenario in the selected countries and the experience so far in dealing with the condition. This is a survey-based study; hence no medications or other treatments will be provided to participants as a part of this study.

ELIGIBILITY:
Inclusion Criteria:

For Experienced/Senior Treating Physicians

* Experienced/senior haematologist treating haemophilia (adult or paediatric) or physician treating patients with haemophilia. (PWH), with greater than 5 years of experience.
* Able to communicate in English or country specific language.
* Agree/sign informed consent before data collection. For Patients Organisations
* Patient organisation supporting haemophilia.
* Expert having greater than 3 years of work experience with the patient organisation.
* Expert level understanding of haemophilia landscape and care pathway in the relevant country.
* Able to communicate in English or country specific language.
* Agree/sign informed consent before data collection. For Patients/Caregivers

  1. Patients of all age groups, diagnosed with haemophilia A or haemophilia B (with or without inhibitors) for greater than 2 years.
  2. For patients less than 18 years of age (*less than 19 years for South Korea), their caregivers aged greater than or equal to 18 years (*greater than or equal to19 years for South Korea) should sign the informed consent.

     *For South Korea, the adult age is 19 years.
  3. Able to communicate in English or country specific language.
  4. Agree/sign informed consent before data collection.

     Exclusion Criteria:
* There is no explicit exclusion criterion in this study, thus any participants group who answers "no" to any of the inclusion criteria will be excluded from the study.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study will enroll 3 types of participant categories:
  1. Experienced/senior treating physicians i.e., haematologists, paediatric haematologist and physicians treating patients with haemophilia (PWH)
  2. Patient organisations (representatives of patient organisations), defined as the organisations working closely to support PWH at a national/regional level
  3. Patients/caregivers.
Sampling Method: Non-Probability Sample
Enrollment: 244 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2025-12-19 (Estimated); Study Completion 2025-12-19 (Estimated)

PRIMARY OUTCOMES:
Estimated prevalence of haemophilia | From start of data collection to end of data collection (approximately 5 months)
  Proportion [%] of individuals in a population
Estimated incidence of haemophilia | From start of data collection to end of data collection (approximately 5 months)
  Number of new cases of haemophilia
Estimated proportion of patients with haemophilia (PWH) who develop inhibitors (%) | From start of data collection to end of data collection (approximately 5 months)
  proportion [%] of individuals in a population

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (4):
- Novo Nordisk Investigational Site, Bangalore, Karnataka, India
- Novo Nordisk Investigational Site, Kuala Lumpur, Malaysia
- Novo Nordisk Investigational Site, Seoul, South Korea
- Novo Nordisk Investigational Site, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com